CLINICAL TRIAL: NCT07150221
Title: Post-Market Clinical Follow-Up Study of the Vivacit-E Vitamin E Highly Crosslinked Polyethylene HXLPE Elevated Liners in Primary THA- A Retrospective Enrollment/Prospective Follow-Up Study
Brief Title: MDR Vivacit-E Elevated Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: MDRG2017-89MS-106H
Record Dates: First submitted 2025-07-29; First posted 2025-09-02 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthritis (OA) of the Hip; Avascular Necrosis of Bone of Hip; Protrusio Acetabuli; Traumatic Arthropathy-Hip; Slipped Capital Femoral Epiphyses; Fused Hip; Fracture of Pelvis; Diastrophic Variant
MeSH Terms: conditions — Osteoarthritis; Slipped Capital Femoral Epiphyses; Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Vivacit-E Elevated Liners: Patients previously implanted with Vivacit-E Elevated Liners.
  Interventions: Device: Vivacit-E Elevated Liners

INTERVENTIONS:
Device: Vivacit-E Elevated Liners — Primary total hip arthroplasty

SUMMARY:
The main objective of this study is to confirm long-term safety, performance, and clinical benefits of the Vivacit-E Vitamin E HXLPE Elevated Liners when used in primary total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patient was 18 years of age or older and skeletally mature at the time of surgery
* Patient qualified for and underwent surgical procedure with a Vivacit-E Vitamin E HXLPE Elevated Liner to treat one of the following indications in primary THA:
* Noninflammatory degenerative joint disease including osteoarthritis and avascular necrosis
* Protrusio acetabuli
* Traumatic arthritis
* Slipped capital epiphysis
* Fused hip
* Fracture of the pelvis
* Diastrophic variant
* Patient underwent surgical procedure 10 years (+ no maximum/- 182 days) prior to date of study consent
* Patient is will and able to sign IRB approved Informed Consent Form or provide verbal consent

Exclusion Criteria:

* Off label use or not according to the approved IFU at the time of surgery
* Patient presented with any of the following at the time of the surgical procedure:
* Osteoradionecrosis
* Neuromuscular compromise, vascular deficiency or other conditions in the affected limb that may lead to inadequate skeletal fixation
* Systemic or local infection
* Revision procedure where other treatment or devices have failed*
* Patient has a psychiatric illness or cognitive deficit that will not allow for proper informed consent
* Uncooperative patient or patient with neurologic disorders who is incapable or unwilling to follow directions

  * For the purpose of this clinical study; a revision procedure refers to a procedure in which the prior procedure on the ipsilateral hip utilized a similar approach (i.e., primary total hip arthoplasty)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population should consist of a maximum of 52 subjects implanted 10 years ago with the Vivacit-E Vitamin E HXLPE Elevated Liner in total hip arthroplasty, according to the approved indications.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Survival of the Implant System via Adverse Events | 10 years
  The primary endpoint is defined by the survival of the implant system at 10 years post-operative, which is based on removal of the study device and will be determined using the Kaplan Meier method. The safety of the study device will be assessed by monitoring the frequency and incidence of adverse events.

SECONDARY OUTCOMES:
Pain and functional performance measured by the Oxford Hip Score | 10 years
  The Oxford Hip Score measures pain and function together, reflecting how hip symptoms impact a patient's severity and frequency of hip-related pain and their physical capabilities.
Subject quality-of-life measured by the EQ-5D-5L | 10 Years
  The EQ-5D-5L is a standardized questionnaire that measures health-related quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. It provides an overall assessment of a participant's perceived health status.

CONTACTS AND LOCATIONS:
Locations (1):
- South Bend Orthopaedics, South Bend, Indiana, United States